CLINICAL TRIAL: NCT03498898
Title: The Effect of Ongoing Beta-blockers Administration on Analgesic Requirements in the Immediate Perioperative Period.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TASMC-17-IM-0598-CTIL
Record Dates: First submitted 2018-04-08; First posted 2018-04-17 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-04

CONDITIONS: Nociceptive Pain
Keywords: Beta adrenergic receptor blockers; Analgesia nociceptive index; Total hip replacement; Total knee replacement
MeSH Terms: conditions — Nociceptive Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A (Active Comparator): American Society of Anesthesiologists (ASA) Score 2-3 with chronic use of Beta adrenergic receptor blockers planned to undergo total hip replacement
  Interventions: Other: Chronic use of Beta adrenergic receptor blocker
- Group B (No Intervention): American Society of Anesthesiologists (ASA) Score 2-3 with no chronic use of Beta adrenergic receptor blockers planned to undergo total hip replacement
- Group C (Active Comparator): American Society of Anesthesiologists (ASA) Score 2-3 with chronic use of Beta adrenergic receptor blockers planned to undergo total knee replacement.
  Interventions: Other: Chronic use of Beta adrenergic receptor blocker
- Group D (No Intervention): American Society of Anesthesiologists (ASA) Score 2-3 with no chronic use of Beta adrenergic receptor blockers planned to undergo total knee replacement

INTERVENTIONS:
Other: Chronic use of Beta adrenergic receptor blocker — Chronic use of Beta adrenergic receptor blocker
  Arms: Group A; Group C

SUMMARY:
This study is designed to discover if chronic use of Beta adrenergic receptor blockers affects pain sensation during and after an elective procedure of hip or knee replacement. The study's population will be divided to four groups: Group A- chronic use of Beta adrenergic receptor blockers undergoing total hip replacement, Group B- no use of Beta adrenergic receptor blockers undergoing total hip replacement, Group C- chronic use of Beta adrenergic receptor blockers undergoing total knee replacement and Group D- no use of Beta adrenergic receptor blockers undergoing total knee replacement. Each patient will be anesthetized using the same anesthesia protocol with pain assessment done by the ANI device intra operatively and by NRS score postoperatively.

DETAILED DESCRIPTION:
The effect of ongoing Beta adrenergic receptor blockers administration on perioperative and post-operative pain.

Beta adrenergic receptor blockers are in common use for treatment of a variety of illnesses. Mostly ones that are connected to the cardiovascular system (such as congestive heart failure, angina pectoris and dysrhythmias) but also for treatment of some neurological disorders and more.

Esmolol and Labetalol are frequently utilized during the perioperative period because of their beneficial effects in treating the acute hemodynamic response to surgical stress. However, clinical studies have confirmed that these adjuvant drugs can reduce postoperative opioid consumption and facilitate earlier extubation. In multiple studies, Esmolol was found effective reducing postoperative pain and the need for narcotic analgesics following surgery. A Meta-analysis published in 2015 in the Journal of Anesthesiology found that Esmolol caused a 32-50% reduction in the need for rescue analgesics and that propranolol decreased the need for rescue analgesics by 72%.

The "Analgesia Nociception Index" (ANI; MetroDoloris Medical Systems, Lille, France), derived from an electrocardiogram (ECG) trace, has been proposed as a noninvasive guide to analgesia. The ANI monitor calculates heart rate variation with respiration, a response mediated primarily by changes in the parasympathetic nervous system (PNS) stimulation to the sinoatrial node of the heart . A painful stimulus will cause a relative decrease in parasympathetic tone and therefore result in a decrease in ANI scores. A score of 100 indicates maximum parasympathetic tone and low nociceptive levels, while a score of zero indicates minimum parasympathetic tone and high nociceptive levels. ANI has been validated in a few studies. In a recently published clinical trial comparing ANI to other predictive modalities and to traditional clinical signs (heart rate and mean arterial pressure) ANI was found to have the highest sensitivity and specificity (P k -0.98) for detecting painful stimulations.

The NRS for pain is a unidimensional measure of pain intensity in adults. The most commonly used is the 11-item NRS which is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0 -10 integers) that best reflects the intensity of their pain where 0 is described as no pain and 10 is described as the worst pain imaginable. The NRS-11 is perhaps the most commonly used pain intensity rating tool with a highly correlated validity to the visual analogue scale (VAS). In addition High test-retest reliability has been observed in both literate and illiterate patients with rheumatoid arthritis (r 0.96 and 0.95, respectively).

ELIGIBILITY:
Inclusion Criteria:

- Candidates for an elective hip replacement.

Exclusion Criteria:

* Patients with no sinus rhythm.
* Patients with an internal cardiac device / cardiac pacemaker.
* The use of Anti muscarinic, alpha adrenergic receptor blockers or anti arhythmic medications.
* Chronic use of Opioids (defined as 20 mg or more of Oxycodone per day for a period of 6 weeks or more).
* BMI> 40.
* Sensitivity to one of the following drugs: Propofol, Fentanyl, Rocuronium, Isoflurane, Morphine, Acetaminophen, Ondansetron.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Fentanyl consumption during surgery. | Intra operative (anaesthesia start until anaesthesia end).
  Measuring the effect of chronic use of Beta adrenergic receptor blockers on the amount of analgesia (Fentanyl).

SECONDARY OUTCOMES:
Post operative Morphine consumption. | Immediate post operative time (from admission to release from PACU).
  Measuring the effect of chronic use of Beta adrenergic receptor blockers on the amount of analgesia (Morphine).
Post operative non opioid analgesia consumption. | Immediate post operative time (from admission to release from PACU).
  Measuring the effect of chronic use of Beta adrenergic receptor blockers on the amount of non opioid analgesia.
Post operative pain (NRS score). | 15 minutes after admission to PACU.
  Measuring the effect of chronic use of Beta adrenergic receptor blockers on NRS pain score.

CONTACTS AND LOCATIONS:
Overall Officials: Idit Matot, MD, PhD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] White PF. What are the advantages of non-opioid analgesic techniques in the management of acute and chronic pain? Expert Opin Pharmacother. 2017 Mar;18(4):329-333. doi: 10.1080/14656566.2017.1289176. Epub 2017 Feb 20. No abstract available. PMID 28132576
- [Background] Chia YY, Chan MH, Ko NH, Liu K. Role of beta-blockade in anaesthesia and postoperative pain management after hysterectomy. Br J Anaesth. 2004 Dec;93(6):799-805. doi: 10.1093/bja/aeh268. Epub 2004 Sep 17. PMID 15377583
- [Background] Collard V, Mistraletti G, Taqi A, Asenjo JF, Feldman LS, Fried GM, Carli F. Intraoperative esmolol infusion in the absence of opioids spares postoperative fentanyl in patients undergoing ambulatory laparoscopic cholecystectomy. Anesth Analg. 2007 Nov;105(5):1255-62, table of contents. doi: 10.1213/01.ane.0000282822.07437.02. PMID 17959952
- [Background] Lopez-Alvarez S, Mayo-Moldes M, Zaballos M, Iglesias BG, Blanco-Davila R. Esmolol versus ketamine-remifentanil combination for early postoperative analgesia after laparoscopic cholecystectomy: a randomized controlled trial. Can J Anaesth. 2012 May;59(5):442-8. doi: 10.1007/s12630-012-9684-x. Epub 2012 Mar 2. PMID 22383085
- [Background] Harkanen L, Halonen J, Selander T, Kokki H. Beta-adrenergic antagonists during general anesthesia reduced postoperative pain: a systematic review and a meta-analysis of randomized controlled trials. J Anesth. 2015 Dec;29(6):934-43. doi: 10.1007/s00540-015-2041-9. Epub 2015 Jul 10. PMID 26160590
- [Background] Funcke S, Sauerlaender S, Pinnschmidt HO, Saugel B, Bremer K, Reuter DA, Nitzschke R. Validation of Innovative Techniques for Monitoring Nociception during General Anesthesia: A Clinical Study Using Tetanic and Intracutaneous Electrical Stimulation. Anesthesiology. 2017 Aug;127(2):272-283. doi: 10.1097/ALN.0000000000001670. PMID 28489614
- [Background] De Jonckheere J, Logier R, Jounwaz R, Vidal R, Jeanne M. From pain to stress evaluation using heart rate variability analysis: development of an evaluation platform. Annu Int Conf IEEE Eng Med Biol Soc. 2010;2010:3852-5. doi: 10.1109/IEMBS.2010.5627661. PMID 21097068
- [Background] Logier R, Jeanne M, De Jonckheere J, Dassonneville A, Delecroix M, Tavernier B. PhysioDoloris: a monitoring device for analgesia / nociception balance evaluation using heart rate variability analysis. Annu Int Conf IEEE Eng Med Biol Soc. 2010;2010:1194-7. doi: 10.1109/IEMBS.2010.5625971. PMID 21095676
- [Background] Upton HD, Ludbrook GL, Wing A, Sleigh JW. Intraoperative "Analgesia Nociception Index"-Guided Fentanyl Administration During Sevoflurane Anesthesia in Lumbar Discectomy and Laminectomy: A Randomized Clinical Trial. Anesth Analg. 2017 Jul;125(1):81-90. doi: 10.1213/ANE.0000000000001984. PMID 28598927
- [Background] Dundar N, Kus A, Gurkan Y, Toker K, Solak M. Analgesia nociception index (ani) monitoring in patients with thoracic paravertebral block: a randomized controlled study. J Clin Monit Comput. 2018 Jun;32(3):481-486. doi: 10.1007/s10877-017-0036-9. Epub 2017 Jun 19. PMID 28631050
- [Background] Jensen MP, McFarland CA. Increasing the reliability and validity of pain intensity measurement in chronic pain patients. Pain. 1993 Nov;55(2):195-203. doi: 10.1016/0304-3959(93)90148-I. PMID 8309709
- [Background] Andersson V, Bergman S, Henoch I, Ene KW, Otterstrom-Rydberg E, Simonsson H, Ahlberg K. Pain and pain management in hospitalized patients before and after an intervention. Scand J Pain. 2017 Apr;15:22-29. doi: 10.1016/j.sjpain.2016.11.006. Epub 2016 Dec 9. PMID 28850341
- [Background] Gruenewald M, Ilies C, Herz J, Schoenherr T, Fudickar A, Hocker J, Bein B. Influence of nociceptive stimulation on analgesia nociception index (ANI) during propofol-remifentanil anaesthesia. Br J Anaesth. 2013 Jun;110(6):1024-30. doi: 10.1093/bja/aet019. Epub 2013 Mar 6. PMID 23471754